CLINICAL TRIAL: NCT07258693
Title: Multimodal Treatment of Knee Osteoarthritis: Comparison of the Combination of Therapeutic Exercise and Noninvasive Neuromodulation (NESA) Versus Therapeutic Exercise and Transcutaneous Electrical Nerve Stimulation (TENS) on Pain, Function, and Mental Health in People Over 60 Years of Age.
Brief Title: Multimodal Treatment of Knee Osteoarthritis: Therapeutic Exercise and Noninvasive Neuromodulation (NESA) Versus Therapeutic Exercise and Transcutaneous Electrical Nerve Stimulation (TENS) in People Over 60 Years of Age.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Responsible Party: Principal Investigator, Agustín Aibar Almazán, Principal investigator, University of Jaén
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: -UUJA
Record Dates: First submitted 2025-11-20; First posted 2025-12-02 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Osteo Arthritis Knee
MeSH Terms: interventions — Exercise Therapy; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise + NESA (Experimental): A treatment group will be enrolled, following an initial assessment and with their consent, in a therapeutic exercise program combined with noninvasive neuromodulation (NESA). The intervention will last 8 weeks. The therapeutic exercise program will consist of 24 sessions, delivered three times a week with supervision, lasting 45-50 minutes per session. In addition, 24 noninvasive neuromodulation (NESA) sessions, each lasting 45 minutes, will be delivered three times a week over the course of the 8 weeks. The main exercise program will include strength, power, balance, and proprioception exercises. The loads will be individualized for each patient, adapting to their accepted pain threshold, physical characteristics, clinical stage, and symptoms. Progression criteria will be established to achieve progressive overload, modifying variables such as repetitions, external load, and range of motion.
  Interventions: Other: Therapeutic exercise and NESA VS. Therapeutic exercise and TENS
- Exercise + TENS (Experimental): A treatment group will receive the same therapeutic exercise program as the experimental group, along with transcutaneous electrical nerve stimulation (TENS). The intervention will last 8 weeks. The therapeutic exercise program will consist of 24 sessions, delivered three times a week with supervision, lasting 45-50 minutes per session. Additionally, 24 sessions of transcutaneous electrical nerve stimulation (TENS) will be delivered three times a week, lasting 45 minutes, distributed over the 8 weeks. The main exercise program will include strength, power, balance, and proprioception exercises. The loads will be individualized for each patient, adapting to their accepted pain threshold, physical characteristics, clinical stage, and symptoms. Progression criteria will be established to achieve progressive overload, modifying variables such as repetitions, external load, and range of motion.
  Interventions: Other: Therapeutic exercise and NESA VS. Therapeutic exercise and TENS

INTERVENTIONS:
Other: Therapeutic exercise and NESA VS. Therapeutic exercise and TENS — The study will include two treatment groups over an 8-week intervention. Group 1 will follow a therapeutic exercise program of 24 supervised sessions (three per week, 45-50 minutes each) combined with 24 sessions of non-invasive neuromodulation (NESA). Group 2 will perform the same therapeutic exercise program but combined with 24 sessions of transcutaneous electrical nerve stimulation (TENS), also delivered three times per week for 45 minutes. The exercise program will include strength, power, balance, and proprioception training, with loads individualized according to pain tolerance, physical condition, clinical phase, and symptoms, and progressed gradually by adjusting repetitions, external load, or range of motion. All participants will be assessed before and after the intervention period, with results recorded systematically.

SUMMARY:
To analyze the effects of therapeutic exercise combined with noninvasive neuromodulation (NESA) or transcutaneous electrical nerve stimulation (TENS) on improving clinical symptoms such as joint pain and stiffness, as well as its impact on the functionality, mental health, and quality of life of people over 60 years of age with knee osteoarthritis.

DETAILED DESCRIPTION:
A single-blind, randomized clinical trial with two intervention groups will be conducted. A pretest-posttest design will be used to evaluate individuals over 60 years of age. Participants will be divided into two groups: one group will receive an 8-week therapeutic exercise program combined with noninvasive neuromodulation (NESA); and the other group will receive the same therapeutic exercise program combined with transcutaneous electrical nerve stimulation (TENS) for 8 weeks. Variables will be measured for both groups using the same validated tools and by the same researchers to avoid information bias and differential misclassification. Assessments will be conducted at the beginning of the intervention and immediately after its completion. The results will be recorded in a database for analysis.

For the independent variables, sociodemographic characteristics will be taken into account. The outcome variables will be divided by domain; pain will be assessed using the Numerical Pain Rating Scale (NPRS), which measures pain intensity. To assess the symptoms and functional capacity associated with knee osteoarthritis, the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) will be used.

For the physical and functional assessment, the Timed Up and Go Test (TUG) will be used to assess functional mobility, balance, and agility. The Short Physical Performance Battery (SPPB) will be used to evaluate balance, gait, and strength/endurance. Balance and gait will also be assessed using the Tinetti Scale. Knee mobility will be measured with a mobile goniometry/inclinometer in flexion and extension. For strength, a dynamometer will be used to measure isometric strength of major knee movements.

Among the psychosocial factors, catastrophizing will be measured with the PCS (Pain Catastrophizing) and kinesiophobia with the abbreviated version of the TSK-11 (Tampa Scale for Kinesiophobia). Fear of falling will be assessed using the Falls Efficacy Scale-International (FES-I).

Quality of life will be measured using the Knee and Hip Osteoarthritis Quality of Life (OAKHQOL) questionnaire. Sleep quality will be measured using the Pittsburgh Index. The Hospital Anxiety and Depression Scale (HADS) will be used for anxiety and depression. Autonomic regulation will be assessed using heart rate variability.

All variables will be measured pre- and post-intervention. As a result, a multimodal treatment is expected to significantly improve clinical symptoms associated with knee osteoarthritis, especially joint pain and stiffness. Additionally, the effectiveness of noninvasive neuromodulation (NESA) will be compared with transcutaneous electrical nerve stimulation (TENS), both in combination with therapeutic exercise. It is also expected to improve functionality, mental health, quality of life, and associated psychosocial factors in people over 60 years of age with knee osteoarthritis. Once the intervention is completed, a final evaluation will be conducted, and the comparative process will determine whether there are significant differences compared to the initial results.

ELIGIBILITY:
Inclusion Criteria:

* Individuals over 60 years of age.
* Diagnosis of knee osteoarthritis in at least one knee according to the clinical criteria of the American College of Rheumatology.
* Ability to walk independently without the need for assistive devices.
* No medical contraindications to physical exercise or the application of noninvasive neuromodulation (NESA).
* Ability to understand and sign the informed consent form to participate in the study.

Exclusion Criteria:

* Present medical contraindications to physical exercise or the application of noninvasive neuromodulation (NSA) (pacemaker, epilepsy, internal bleeding, acute febrile processes, acute thrombophlebitis, and/or phobia of electricity).
* Present active oncological diseases or systemic autoimmune diseases.
* Present severe psychiatric or neurological disorders that limit understanding and collaboration in treatment.
* History of any surgery or fracture of the affected lower limb in the last 3 months.
* Presence of severe gait or balance difficulties that impede the performance of the proposed exercises.
* Simultaneous participation in other clinical trials.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2026-01-07 (Estimated); Primary Completion 2026-01-12 (Estimated); Study Completion 2026-04-07 (Estimated)

PRIMARY OUTCOMES:
Pain Score - Numeric Rating Scale for Pain (0-10) | Up to eight weeks
  Pain intensity will be assessed using the Numeric Rating Scale for Pain, which ranges from 0 to 10, where 0 indicates no pain and 10 represents the worst pain imaginable. A reduction of ≥2 points is considered clinically significant.
Western Ontario and McMaster Universities Osteoarthritis Index | Up to eight weeks
  Knee osteoarthritis symptoms will be assessed using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), which evaluates pain, stiffness, and physical function. Higher scores indicate worse symptoms.
Knee Range of Motion - Goniometer | Up to eight weeks
  Knee joint range of motion will be evaluated using a goniometer. Lower values indicate reduced mobility, commonly associated with disease severity.
Strength Tests - Hand-held Dynamometry | Up to eight weeks
  Isometric muscle strength of the quadriceps, hamstrings, and handgrip will be measured using a hand-held dynamometer, expressed in kilograms (kg) or newtons (N). Lower scores indicate muscle weakness, often linked to osteoarthritis progression.
Timed Up and Go (TUG) Performance | Up to eight weeks
  Functional mobility will be assessed using the Timed Up and Go test, measured in seconds (standing up, walking 3 m, turning, and sitting down). Values >12 seconds indicate an increased risk of falls.
Short Physical Performance Battery - Global Score | Up to eight weeks
  Physical performance will be assessed through balance tests, gait speed, and sit-to-stand tasks. Scores ≤9 indicate functional limitation.
Tinetti Balance and Gait Score | Up to eight weeks
  Balance and gait will be evaluated using the Tinetti Assessment Tool, ranging from 0 to 28, where scores <19 indicate a high risk of falls.
Pain Catastrophizing Scale. | Up to eight weeks
  Pain catastrophizing will be assessed with the Pain Catastrophizing Scale, ranging from 0 to 52. Scores ≥30 indicate clinically relevant catastrophizing.
Total TSK-11 Score - Tampa Scale for Kinesiophobia | Up to eight weeks
  Kinesiophobia will be measured using the 11-item Tampa Scale for Kinesiophobia, with scores ranging from 11 to 44. Scores ≥23 indicate high fear of movement.
Falls Efficacy Scale-International | Up to eight weeks
  Fear of falling will be assessed using the FES-I, ranging from 16 to 64. Scores >23 indicate concern, and >28 indicate high concern about falling.
Pittsburgh Sleep Quality Index | Up to eight weeks
  Sleep quality will be assessed using the Pittsburgh Sleep Quality Index, which ranges from 0 to 21, with scores >5 indicating poor sleep quality.
Osteoarthritis Knee and Hip Quality of Life Questionnaire | Up to eight weeks
  Quality of life will be evaluated using the Osteoarthritis Knee and Hip Quality of Life Questionnaire, covering physical, mental, and social domains. Higher scores reflect greater impairment.
Hospital Anxiety and Depression Scale | Up to eight weeks
  Anxiety and depression will be evaluated using the Hospital Anxiety and Depression Scale, with each subscale ranging from 0 to 21. Scores ≥11 indicate clinically significant symptoms.
Heart Rate Variability Parameters | Up to eight weeks
  Autonomic regulation will be assessed through heart rate variability parameters (SDNN, RMSSD, LF/HF ratio) using ECG or a validated wearable device. Lower HRV indicates poorer autonomic regulation.

CONTACTS AND LOCATIONS:
Locations (1):
- ICOT rehabilitation centers, Las Palmas de Gran Canaria, Spain